CLINICAL TRIAL: NCT01004913
Title: Evaluation of the Otolithic Organs Function in Patients Suffering From Benign Paroxysmal Positional Vertigo (BPPV) by Vestibular Evoked Myogenic Potentials (VEMP).
Brief Title: Vestibular Evoked Myogenic Potentials in Benign Paroxysmal Positional Vertigo (VEMP in BPPV)
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other)
Responsible Party: Sponsor
Other Study IDs: kehila106/109
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2011-08

CONDITIONS: Vertigo
Keywords: Benign paroxysmal positional vertigo; Vestibular evoked myogenic potentials; Sacculo-colic reflex
MeSH Terms: conditions — Vertigo; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is the most frequent cause of vertigo of peripheral vestibular origin with life time incidence of 2.4%. BPPV is characterized by bouts of acute whirling vertigo lasting less than one minute provoked by changes in head position in relation to the gravitational vector. The vertigo is accompanied by typical rotational or horizontal nystagmus that is often demonstrated by the Dix-Hallpike maneuver and less frequently by testing for positional nystagmus. BPPV pathogenesis is currently explained by the fall of otoconia (calcium-carbonate crystals) or otoconial debris from the tectorial membrane of the otolithic organs into the dependant semicircular canals (canalithiasis) or adherence of such particles to the semicircular canal's cupula (cupulithiasis). Under these circumstances, the semicircular canal which normally responds only to angular velocity and acceleration is stimulated by gravity. Otoconial remnants as free floating particles inside the semicircular canal arms or attached to the cupula have been observed by few investigators. Although the presence of such particles explains most characteristics of the positioning nystagmus described in BPPV, it does not account for the dizziness and disequilibrium which are described by many patients even without changes in head position and the continuation of such symptoms after successful treatment of BPPV as evidenced by the resolution of positional vertigo and nystagmus.

The study hypothesis is that otolithic pathology is an important component in the pathogenesis of BPPV explaining these symptoms, BPPV recurrence, and the refractoriness of some BPPV cases to the vastly employed particles repositioning treatments. In the present study the Vestibular Evoked Myogenic Potentials (VEMP) testing would be employed to measure the function of one of the otolithic organs - the saccule. The study objectives are: 1. To investigate possible malfunction of the saccule in patients suffering from BPPV. 2. To look for association between saccular pathology and BPPV recurrence and between such pathology and BPPV treatment failure. 3. To study possible relation between saccular pathology and continuation of dizziness and disequilibrium despite the resolution of positional vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Complaints of positional or positioning vertigo.
* Presence of typical nystagmus for posterior canal BPPV in Dix Hallpike maneuver

Exclusion Criteria:

* Patient younger than 18 or older than 60 years of age.
* Otoneurology bed-side examination reveals bilateral BPPV.
* Audiometry and tympanometry show conductive hearing loss.
* Signs of retrocochlear lesion or central vestibular pathology in bed-side otoneurological examination or audiometry or ENG/VNG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering fron Benign Paroxysmal Positional Vertigo
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with normal VEMP response | At the time of diagnosis of BPPV

SECONDARY OUTCOMES:
Number of subjects with recurrent BPPV in whom VEMP response was pathological | at the time of BPPV diagnosis

OTHER OUTCOMES:
no other outcome measures | no other outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Otoneurology Unit, Lin Medical Center, 35 Rotchild Avenue, Haifa, Israel

REFERENCES:
- [Derived] Shupak A, Falah R, Kaminer M. Functional Integrity of the Inferior Vestibular Nerve and Posterior Canal BPPV. Front Neurol. 2020 Aug 26;11:894. doi: 10.3389/fneur.2020.00894. eCollection 2020. PMID 32982924